CLINICAL TRIAL: NCT03798158
Title: Prevalence and Characterization of Persistent Dyspnea After an Hospitalization for a Respiratory Disease
Brief Title: Prevalence and Characterization of Persistent Dyspnea After Hospitalization
Acronym: DyHP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02757-48
Record Dates: First submitted 2018-11-21; First posted 2019-01-09 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Dyspnea; Pulmonary Disease
MeSH Terms: conditions — Dyspnea; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multidisciplinary Dyspnea Profile questionnaire — Multidisciplinary Dyspnea Profile questionnaire at the beginning and the end of an hospitalization

SUMMARY:
The investigators aim to make an overview of persistent dyspnea at the end of an hospitalization for a respiratory disease using an actual tool, the Multidisciplinary Dyspnea Profile questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Able to respond the questionnaire
* Presenting at admission a dyspnea over 3/10 on numerical analogic scale
* Admitted for a respiratory cause

Exclusion Criteria:

* cognitive impairment
* aphasia
* no french-speaking person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every consecutive patient admitted to hospitalization for a respiratory cause having a significant dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of persistent dyspnea in the end of an hospitalization for a a respiratory disease | An average of one week, until the end of the hospitalization

SECONDARY OUTCOMES:
Characterization of persistent dyspnea using MDP | An average of one week, until the end of the hospitalization
Outcome of patients with persistent dyspnea after hospitalization | 6 months
  6 months mortality, incidence of rehospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- ADOREPS, Paris, France